CLINICAL TRIAL: NCT01228448
Title: Pilot Study of In-Room PET in Proton Radiation Therapy
Brief Title: In-Room PET in Proton Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Helen A. Shih, MD, Attending Radiation Oncologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-241
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Brain Tumor; Head and Neck Tumor; Skull Base Tumor
Keywords: external beam proton radiotherapy; PET
MeSH Terms: conditions — Brain Neoplasms; Head and Neck Neoplasms; Skull Base Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Participants 1-39 (Experimental): PET Scan done right after one radiation treatment is complete and will take 15-20 minutes. After undergoing their first PET scan, participants will have the option to undergo 1-2 additional scans throughout radiation treatment in the same manner as the first scan.
  Interventions: Procedure: PET scan

INTERVENTIONS:
Procedure: PET scan — In-Room PET scan

SUMMARY:
The investigational part of this study is using a mobile PET/CT scanner to take images of the participants tumor immediately after they are treated with proton radiation. This allows the participant to be treated and imaged on the same bed. The information obtained may improve the accuracy of treatment and may help to minimize the dose delivered unnecessarily to healthy tissue.

DETAILED DESCRIPTION:
For all participants, right after one regular treatment fraction, NeuroPET or NeuroPET II will be wheeled into the patient room. The patient bed will be moved directly into the scan position and a PET scan will be acquired in list-mode for 15 to 20 minutes followed by a CT scan for ~5 minutes. After undergoing their first PET scan, participants will have the option to undergo 1-2 additional scans throughout radiation treatment in the same manner as the first scan.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with brain, head and neck, and skull base tumors receiving external beam proton radiotherapy at the Francis H. Burr Proton Therapy Center at MGH
* Age 18 or over
* ECOG Performance status 0, 1 or 2

Exclusion Criteria:

* Uncontrolled intercurrent illness that, in the opinion of the investigator, would limit the participant's compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-10; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness | 2 years
  Acquire PET/CT scan data in list-mode on patients undergoing external beam proton radiotherapy for brain and soft tissue tumors in head. Analyze these data to assess the effectiveness of using PET/CT for in-room PET monitoring for proton radiation therapy quality assurance.

SECONDARY OUTCOMES:
Optimize the in-room PET acquisition length | 2 years
  Reconstruct these list-mode PET data for different scan durations and optimize in-room PET acquisition length

CONTACTS AND LOCATIONS:
Overall Officials: Helen A. Shih, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States